CLINICAL TRIAL: NCT06019494
Title: Is Flow Rate During Oocyte Retrieval Associated With the Number of Oocytes Retrieved? A Randomized Control Trial
Brief Title: Comparison of 2 Different Flow Rates During Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eugonia (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Flow rate for oocyte retrieval
Record Dates: First submitted 2023-08-08; First posted 2023-08-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Infertility
Keywords: Flow rate; Aspiration pressure; Oocyte retrieval
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low aspiration flow rate (Experimental): All follicles will be aspirated with the addition of follicular flushing if necessary with an aspiration flow rate of 0.42ml/sec.
  Interventions: Procedure: Oocyte retrieval with low aspiration flow rate
- High aspiration flow rate (Experimental): All follicles will be aspirated with the addition of follicular flushing if necessary with an aspiration flow rate of 0.62ml/sec.
  Interventions: Procedure: Oocyte retrieval with high aspiration flow rate

INTERVENTIONS:
Procedure: Oocyte retrieval with low aspiration flow rate — All follicles will be aspirated with the addition of follicular flushing if necessary (up to 5 times per follicle) with an aspiration flow rate of 0.42 ml/sec.
  Arms: Low aspiration flow rate
Procedure: Oocyte retrieval with high aspiration flow rate — High aspiration flow rate All follicles will be aspirated with the addition of follicular flushing if necessary (up to 5 times per follicle) with an aspiration flow rate of 0.62 ml/sec.
  Arms: High aspiration flow rate

SUMMARY:
The purpose of this study is to evaluate the effect of different flow rates during oocyte retrieval, on the number of cumulus oocyte complexes (COCs) retrieved.

DETAILED DESCRIPTION:
In the current study, each ovary will be randomly allocated to oocyte retrieval using 0.42 ml/sec or 0.62 ml/sec flow rate.

The primary endpoint will be the number of oocytes retrieved, while secondary outcomes will include oocyte recovery rate (number of oocytes retrieved per follicle aspirated), number of mature oocytes, maturation rate (number of mature oocytes/number of oocytes retrieved), mean oocyte score (by evaluating oocyte shape and size, ooplasm characteristics, structure of perivitelline space (PVS), structure of zona pellucida (ZP) and polar body (PB) morphology), fertilization rate (number of fertilized oocytes/number of mature oocytes), number of blastocysts and blastulation rate (number of blastocysts/number of 2PN).

Patients aged 18-43 years with the presence of at least 3 follicles ≥ 11mm in each ovary on the day of oocyte retrieval will be eligible for inclusion in the study.

Prior to oocyte retrieval in eligible patients their left and right ovary will be randomly allocated into the 0.42 ml/sec or 0.62 ml/sec flow rate group. Randomisation with minimisation will be employed.

The specific flow rates will be achieved by adjusting the aspiration pressure of the vacuum pump accordingly. A study nurse will be responsible for adjusting the aspiration pressure of the vacuum pump depending on randomization. The doctor performing the oocyte retrieval will not be aware of the flow rate used in each ovary.

All follicles will be aspirated and then flushed if needed up to a maximum of 5 times with an open flushing technique, using a 16G double-lumen needle.

Data will be registered regarding the number of flushes required to retrieve a COC, the morphology of oocytes after denudation, oocyte fertilisation and embryo development up to the blastocyst stage.

ELIGIBILITY:
Inclusion Criteria:

* Presence of both ovaries
* 18-43 years old
* At least 3 follicles ≥ 11mm in each ovary on the day of oocyte retrieval

Exclusion Criteria:

* One or no ovaries present
* Monofollicular development
* Poor responders
* Previous history of hemorrhage during oocyte retrieval

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must have both ovaries present
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | During oocyte retrieval
  Number of oocytes retrieved per ovary randomised.

SECONDARY OUTCOMES:
Oocyte recovery rate | During oocyte retrieval
  Number of oocytes retrieved per follicle aspirated.
Oocyte maturation rate | 2-3 hours post oocyte retrieval
  Number of mature (metaphase-II) oocytes divided by the number of oocytes retrieved per ovary randomised.
Average oocyte score | 2-3 hours post oocyte retrieval
  Average oocyte score based on the evaluation of oocyte shape and size, ooplasm characteristics, structure of perivitelline space, structure of zona pellucida and polar body morphology.
Fertilization rate | Day 1 post oocyte retrieval
  Number of fertilised (2PN) oocytes divided by the number of matured oocytes retrieved per ovary randomised.
Percentage of good quality blastocysts on day 5 | 5 days post oocyte retrieval
  Number of good quality blastocysts divided by the number of fertilized oocytes per ovary randomised.

CONTACTS AND LOCATIONS:
Overall Officials: George T Lainas, PhD, Principal Investigator — Eugonia ART Unit
Locations (1):
- Eugonia Unit of Assisted Reproduction, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazzaroni-Tealdi E, Barad DH, Albertini DF, Yu Y, Kushnir VA, Russell H, Wu YG, Gleicher N. Oocyte Scoring Enhances Embryo-Scoring in Predicting Pregnancy Chances with IVF Where It Counts Most. PLoS One. 2015 Dec 2;10(12):e0143632. doi: 10.1371/journal.pone.0143632. eCollection 2015. PMID 26630267